CLINICAL TRIAL: NCT00668473
Title: Endostatin and Other Angiogenic/Angiostatic Mediators in Patients With Systemic Sclerosis
Brief Title: Angiogenic/Angiostatic Mediators in Patients With Systemic Sclerosis
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Kristine Phillips, clinical assistant professor, University of Michigan
Other Study IDs: HUM00011196
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Systemic Sclerosis
Keywords: systemic sclerosis angiogenesis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — skin serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Subjects with diffuse scleroderma
- 2: Healthy controls

SUMMARY:
We propose to examine several angiogenic/angiostatic mediators in the skin and serum of subjects with SSc and compare it to levels found in the skin and serum of healthy subjects.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a connective tissue disease that is characterized by fibrosis of the skin and internal organs. One of the earliest pathologic changes in patients with SSc is damage to the blood vessels. Many abnormalities have been found in the inner layer of the blood vessel, the enothelial tissue. It is known that there are mediators in the blood and tissues of the body that affect the endothelial tissue. These are called angiogenic (promote blood vessel formation) and angiostatic (inhibit blood vessel formation) mediators. Many of these mediators have been examined in the peripheral blood of patients with SSc, but fewer of these mediators have been examined at the site of action, in the tissue near the microvasculature. We hypothesize that there are differences in the levels of angiogenic/angiostatic mediators between healthy subjects and subjects with SSc. In addition, we propose that there are differences at skin sites that have varying levels of involvement with SSc of these angiogenic/angiostatic factors in subjects with SSc.

ELIGIBILITY:
Inclusion Criteria:

1. Meet American College of Rheumatology criteria for systemic sclerosis
2. Subjects with systemic sclerosis must have involvement proximal to the knee or elbow, excluding the face
3. Persons with no chronic health conditions

Exclusion Criteria:

1. Persons with systemic sclerosis as a result of being exposed to chemicals or drugs that can cause a sceroderma-like illness
2. Persons with autoimmune diseases other than systemic sclerosis
3. Persons treated with cyclophosphamide in the last 8 weeks
4. Persons with active infections, including but not limited to hepatitis C, hepatitis B, and HIV
5. Persons prone to bleeding because they are treated with medications that thin the blood or have a low platelet count

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Attendees of a tertiary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-05; Primary Completion 2008-05 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Level of endostatin in skin and serum | At time of of biopsy and blood draw

SECONDARY OUTCOMES:
Level of JAM-A in skin and serum | At time of blood draw and skin biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Phillips, MD, Principal Investigator — University of Michigan; James R Seibold, MD, Principal Investigator — University of Michigan; Alisa E Koch, MD, Principal Investigator — University of Michigan; Julie A Konkle, BSN, Study Director — University of Michigan
Locations (1):
- University of Michigan Hospitals, Ann Arbor, Michigan, United States